CLINICAL TRIAL: NCT00376857
Title: Surgical Removal of Idiopathic Epiretinal Membrane With and Without the Assistance of Indocyanine Green: a Randomised Controlled Clinical Trial
Brief Title: Surgical Removal of Idiopathic Epiretinal Membrane With and Without the Assistance of Indocyanine Green.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regensburg (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03123
Record Dates: First submitted 2006-09-13; First posted 2006-09-15 (Estimated); Last update posted 2006-09-15 (Estimated); Status verified 2006-09

CONDITIONS: Idiopathic Epiretinal Membrane, Cataract
Keywords: Indocyanine green, toxicity, epiretinal membrane, visual field defect
MeSH Terms: conditions — Cataract; Epiretinal Membrane | interventions — Surgical Procedures, Operative

INTERVENTIONS:
Drug: Surgery with and without the aid of Indocyanine Green (ICG)

SUMMARY:
It was the aim of the present study to prospectively compare the functional and morphological outcome of idiopathic epiretinal membrane surgery with and without the assistance of Indocyanine green (ICG). The main outcome measure was improvement of best-corrected visual acuity (BCVA). This was treated as an open question and we had no hypothesis which of the two therapies was superior.

ELIGIBILITY:
Inclusion Criteria:

* Patients with IEM and cataract or posterior chamber intraocular lens pseudophakia complaining of loss of visual acuity and metamorphopsia during the past six months.

Exclusion Criteria:

* Other retinal disease, non-idiopathic epiretinal membrane, glaucoma or history of retinal detachment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60

PRIMARY OUTCOMES:
The main outcome measure was improvement of best-corrected visual acuity (BCVA).

SECONDARY OUTCOMES:
Other outcome measures included postoperative BCVA, status of Amsler grid test, reduction of macular retinal thickness, residual or recurrent macular epiretinal membrane

CONTACTS AND LOCATIONS:
Overall Officials: Jost Hillenkamp, MD, Principal Investigator — Dept. of Ophthalmology, University of Regensburg; Parykshit Saikia, MD, Principal Investigator — Dept. of Ophthalmology, University of Regensburg; Helmut G Sachs, MD, Study Chair — Dept. of Ophthalmology, University of Regensburg
Locations (1):
- Dept. of Ophthalmology, University of Regensburg, Regensburg, Germany

REFERENCES:
- [Derived] Hillenkamp J, Saikia P, Herrmann WA, Framme C, Gabel VP, Sachs HG. Surgical removal of idiopathic epiretinal membrane with or without the assistance of indocyanine green: a randomised controlled clinical trial. Graefes Arch Clin Exp Ophthalmol. 2007 Jul;245(7):973-9. doi: 10.1007/s00417-006-0485-1. Epub 2006 Dec 21. PMID 17186261